CLINICAL TRIAL: NCT03062904
Title: Search of a Paradoxical Fall in Maximum Expiratory Flow After Bronchodilation in Healthy Subjects
Acronym: VACUVOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P120301; 2012-A01643-40 (Other: IDRCB)
Record Dates: First submitted 2017-01-10; First posted 2017-02-24 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2017-10

CONDITIONS: Paradoxical Fall in Maximum Expiratory Flows
Keywords: healthy; respiratory system; ventilation; paradoxical effect; methacholine; bronchodilator; NEP; EFL
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- drug (Experimental)
  Interventions: Drug: Inhaled Bronchodilators +/- Inhaled Methacholine

INTERVENTIONS:
Drug: Inhaled Bronchodilators +/- Inhaled Methacholine — 1. Combined Salbutamol 200μg and Ipratropium bromure 80μg (2 inhalations) if paradoxal answer
  2. Inhaled Methacholine based on international recommendations

SUMMARY:
There exists a physiological limitation of the expiratory flows because of the physical properties of the bronchial tree (flexible bronchial walls in a complex architecture subjected to variations of pressure and volume). For a given lung, in a given state, for each pulmonary volume there is a corresponding Maximum Expiratory Flow (MEF). In healthy subject, the bronchial smooth muscles have a basal tonicity which is not negligible. If the tonicity is increased, this generally leads to a reduction in MEF. If it is decreased, MEF rather tends to increase, there are healthy individuals for whom the inhibition of the contraction of the bronchial smooth muscles by inhalation of bronchodilatator leads to a reduction in the MEF: this is called "paradoxical effect". When this reduction exists, it appears it occurs at low pulmonary volumes (approximately 50% for a volume of less than 25% of the CV). Under this circumstance, it seems that the basal tonicity of the bronchial smooth muscles would fight against the expiratory collapse of the bronchi, and this would happen especially for distal bronchi, for low pulmonary volume and for forceful expiration. The existence of such a phenomenon would be in favour of a "stiffening" role of the bronchial smooth muscles. The bronchial smooth muscles would not be only harmful cells causing of the asthma attacks.

DETAILED DESCRIPTION:
There exists a physiological limitation of the expiratory flows because of the physical properties of the bronchial tree (flexible bronchial walls in a complex architecture subjected to variations of pressure and volume). For a given lung, in a given state, for each pulmonary volume there is a corresponding Maximum Expiratory Flow (MEF). In healthy subject, the bronchial smooth muscles have a basal tonicity which is not negligible. If the tonicity is increased, this generally leads to a reduction in MEF. If it is decreased, MEF rather tends to increase, there are healthy individuals for whom the inhibition of the contraction of the bronchial smooth muscles by inhalation of bronchodilatator leads to a reduction in the MEF: this is called "paradoxical effect". When this reduction exists, it appears it occurs at low pulmonary volumes (approximately 50% for a volume of less than 25% of the CV). Under this circumstance, it seems that the basal tonicity of the bronchial smooth muscles would fight against the expiratory collapse of the bronchi, and this would happen especially for distal bronchi, for low pulmonary volume and for forceful expiration. The existence of such a phenomenon would be in favour of a "stiffening" role of the bronchial smooth muscles. The bronchial smooth muscles would not be only harmful cells causing of the asthma attacks.

Primary end-point:

The aim of this study is to evaluate the occurrence or increase of the Expiratory Flow Limitation (EFL) under either Negative Expiratory Pressure (NEP) or submaximal gentle forced expiratory manoeuvres (partial flow-volume loops at tidal volume) after bronchodilation in certain healthy men breathing at low pulmonary volumes (by applying a chest wall strapping).

Secondary end-point:

The secondary objectives are

* to evaluate the effect of the fall of the tonicity of the bronchial smooth muscles (normal and constrained pulmonary volumes) on the following criteria/variables:

  * the closing volume: we would expect an increase of it.
  * modifications of forced flow-volume loop; we would expect a reduction in the MEF at low lung volumes.
  * some modifications of the Pulmonary Function Test (PFT); we would expect an absence of significant difference in certain pulmonary volumes (Vital Capacity - VC, Total Lung Capacity -TLC,…), perhaps with a reduction in the Inspiratory Capacity (IC), an increase in airways resistances by high frequency oscillation
* Validation of the digital model of expiration of Florens-Filoche: towards a tool of assistance to the interpretation of the PFT.

During the various experimental sessions, we will record a certain "number" of variables that will be necessary to "feed" the final model of Florens-Filoche, such as:

* Oesophageal Pressure, Mouth Pressure: continuously. Static oesophageal pressure at:
* Residual Volume -RV, TLC, VC
* flows and pulmonary volumes continuously.

This study will attempt to develop a tool to assist in the interpretation of the PFT:

* earlier disease detection (of the bronchial smooth muscles),
* better follow-up of obstructive pathologies, their response to the treatment,
* simplification of the diagnosis of asthma,
* automation of interpretation…

Study Design:

The study includes 3 visits, as follows:

Visit 0:

Anthropometric characteristics Medical screening and eligibility criteria Chest X-ray ECG Blood pressure Pulse oximetry, heart rate PFT

Visit 1:

The first visit (V1) will last 3h and 30 minutes roughly and will consist of:

* PFT: spirometry, maximal flow-volume loops (MFVL), in sitting position.
* Closing Volume and airways resistances in sitting position.
* Insertion of a small oesophageal catheter for continuous monitoring of the oesophageal pressure and measurement of static pressure at some volumes
* Thoraco-abdominal (chest wall) strapping
* Measures of slow VC and MFVL in lying position
* Either NEP in lying position or submaximal gentle forced expiratory manoeuvres (partial flow-volume loops at tidal volume)
* Removal of the thoraco-abdominal (chest wall) strapping
* Test of Bronchodilatation (combined Salbutamol 200μg and Ipratropium bromure 80μg; 2 inhalations): wait 30 min and then
* Thoraco-abdominal (chest wall) strapping
* Either NEP or submaximal gentle forced expiratory manoeuvres (partial flow-volume loops at tidal volume)
* Measures of slow VC and MFVL in lying position
* Removal of the thoraco-abdominal (chest wall) strapping
* Measures of slow VC and MFVL in sitting position
* Removal of the small oesophageal catheter
* Closing Volume and airways resistances in sitting position

Each measurement will be repeated at least 3 times, until at least 2 reproducible measurements are obtained.

Visit 2:

The second meeting (V2) will be proposed only to participants who will present with a reduction in some of their MEF at the time of V1 of the protocol. It will consist of Methacholine Challenge Test. The duration of this test is approximately 1 hour.

Number of Subjects to be included: 65 healthy subjects under 35y are necessary find at lest 6 subjects presenting with a "paradoxal effect".

Duration of the study: two years

ELIGIBILITY:
Inclusion Criteria:

All the volunteers will:

* be between 18 and 35 years/old
* be male (because of binding thoracic, more difficult to realize and more uncomfortable in the female subjects)
* have to understand French
* have to be affiliated to the social security
* have to be "non smokers, or having never smoked"
* have to have read and have understood the information record
* have to have signed the informed consent
* have to not to be involved in a former scientific study.
* abnormal PFT (at least one value below the lower limit of normal)
* Abnormal chest radiography
* Abnormal ECG

Exclusion Criteria:

* Chronic pathology
* Long-standing treatments, recent vaccination (< 3 weeks), recent bronchitis (< 3 weeks)
* Cardio-respiratory diseases, in particular: asthma, COPD, previous pneumothorax, hemoptyses, acute coronary syndrome, uncontrolled and/or untreated cardiac arrhythmia, bradycardia (<55bpm), arterial hypertension (diastolic>95mmHg, systolic>150mmHg),
* Current abdominal disease (clinical or known hepatomegaly, irritable bowel syndrome, etc…), gastro-oesophageal reflux
* BMI < 18 and > 26
* Disorder of coagulation (and anticoagulant treatment), frequent epistaxis
* Porphyrae
* Epilepsy, Cerebrovascular accident (stroke or transient ischemic attack) < 3 months
* Severe hepatic Insufficiency
* Glaucoma
* Benign Prostatic Hypertrophy
* Allergy: latex, lidocaine, salbutamol, ipratropium or parasympathomimetic agents
* Current allergic rhino-conjunctivitis
* History of previous oedema of Quincke or anaphylactic shock
* Aneurism of the aorta, cerebral aneurism or another arterial aneurism
* Myasthenia
* Thyroid disorders
* Protected underage child and adults

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Estimated)
Dates: Start 2014-02; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence or increase of the Expiratory Flow Limitation (EFL) under either Negative Expiratory Pressure (NEP) or submaximal gentle forced expiratory manoeuvres (partial flow-volume loops at tidal volume) | After bronchodilation, up to 2 hours
  The aim of this study is to evaluate the occurrence or increase of the Expiratory Flow Limitation (EFL) under either Negative Expiratory Pressure (NEP) or submaximal gentle forced expiratory manoeuvres (partial flow-volume loops at tidal volume) after bronchodilation in certain healthy men breathing at low pulmonary volumes (by applying a chest wall strapping).

SECONDARY OUTCOMES:
Evaluation of the effect of the fall of the tonicity of the bronchial smooth muscles (normal and constrained pulmonary volumes) on the closing volume | after bronchodilation while breathing at low pulmonary volumes (by applying a chest wall strapping), up to 2 hours
Evaluation of the effect of the fall of the tonicity of the bronchial smooth muscles (normal and constrained pulmonary volumes) on the modifications of forced flow-volume loop | after bronchodilation while breathing at low pulmonary volumes (by applying a chest wall strapping), up to 2 hours
Evaluation of the effect of the fall of the tonicity of the bronchial smooth muscles (normal and constrained pulmonary volumes) on the inspiratory capacity airways resistances | after bronchodilation while breathing at low pulmonary volumes (by applying a chest wall strapping), up to 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pierantonio Laveneziana, MCUPH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Pitié-Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No